CLINICAL TRIAL: NCT05915949
Title: Evaluation of the Efficacy of Combination of Dapagliflozin and Lobeglitazone on Glucose Concentrations and Body Fat in Patients With Type 2 Diabetes
Brief Title: Comparison of Dapagliflozin, Lobeglitazone, and Its Combination in Efficacy and Safety
Acronym: Location-F
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1910-568-001
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Type 2
Keywords: diabetes type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; lobeglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg once daily will be given to participants.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Lobeglitazone (Active Comparator): Lobeglitazone 0.5 mg once daily will be given to participants.
  Interventions: Drug: Lobeglitazone 0.5 mg
- Dapagliflozin and Lobeglitazone combined (Active Comparator): Dapagliflozin 10 mg and lobeglitazone 0.5 mg once daily together will be given to participants.
  Interventions: Drug: Dapagliflozin + Lobeglitazone

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Forxiga 10mg Tab once daily will be given to participants for 24 weeks.
  Other Names: Forxiga 10mg
  Arms: Dapagliflozin
Drug: Lobeglitazone 0.5 mg — Duvie 0.5mg Tab once daily will be given to participants for 24 weeks.
  Other Names: Duvie 0.5 mg
  Arms: Lobeglitazone
Drug: Dapagliflozin + Lobeglitazone — Duvie 0.5mg Tab once daily will be given to participants for 24 weeks.
  Other Names: Forxiga 10mg + Duvie 0.5mg
  Arms: Dapagliflozin and Lobeglitazone combined

SUMMARY:
Diabetes is the most frequently occurring chronic disease along with obesity, hypertension, and hyperlipidemia. The number of patients with diabetes is increasing worldwide. Despite rapid progress in management of diabetes, the problem is that glycemic target goal is still low showing 30-40%. Thus, diabetes has become a serious social, economic, and public health problem beyond individual health problems due to its increasing prevalence.

DETAILED DESCRIPTION:
Previously, metformin, sulfonylurea, and insulin injections were used to treat diabetes, but since then, various new drugs such as thiazolidinedione (TZD), sodium-glucose cotransporter-2 (SGLT-2) inhibitor, dipeptidyl peptidase-4 (DPP-4) inhibitor, and glucagon like peptide-1 (GLP-1) receptor agonist have been released. Among them, metformin and TZD are known to improve insulin resistance, SGLT-2 inhibitor has a mechanism to excrete glucose into urine, and other drugs have a mechanism to promote insulin secretion.

After a report in 2007 that rosiglitazone could increase cardiovascular disease, use of TZD has been limited. However, more people are having insulin resistance, and this is more evident in developing countries. In this circumstance, TZD can be a main stay for diabetic patients with insulin resistance. TZDs improve insulin sensitivity by activating peroxisome proliferator-activated receptor γ (PPARγ). They have shown excellent glycemic durability. On the other hand, SGLT-2 inhibitors are attracting attention as a mechanism that directly excretes excess glucose in diabetic patients through urine. Many cardiovascular outcome trials have proven its efficacy in cardiovascular and renal outcomes. Current guidelines proposed a new paradigm in the management of T2DM, with a preferential place for SGLT-2 inhibitors, after metformin, in patients with atherosclerotic cardiovascular disease, heart failure and progressive kidney disease.

As such, combination therapy of TZD and SGLT-2 inhibitors, two drugs that have mechanisms for improving insulin resistance and urinary glucose excretion, would have compensatory effects, which would be effective for diabetes treatment. In addition, since studies that investigated effect of TZD and SGLT-2 inhibitor combination on changes in body fat mass and metabolic phenotype are lacking, we investigated the effect of reducing visceral fat (abdominal visceral fat mass/abdominal subcutaneous fat mass) in combination therapy with dapagliflozin, an SGLT-2 inhibitor, and lobeglitazone, a TZD.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients between the ages of 20 and 80 who are taking oral diabetes medications (metformin and/or DPP-4 inhibitors) for more than 8 weeks without dose adjustment
* body mass index (BMI) ≥ 20 kg/m2
* eGFR ≥ 50 mL/min/1.73 m2
* HbA1c: 7-10%.

Exclusion Criteria:

* patients with type 1 diabetes; HbA1c <7% or HbA1c >10%
* fasting blood glucose (FPG) >15 mmol/L (270 mg/dL) at the first visit (screening) and pre-randomization screening
* women of childbearing potential (if not using proper contraception)
* history of gastric surgery (including gastric banding within 3 years)
* history of diabetic ketoacidosis or non-ketogenic hyperosmotic coma
* average of 3 blood pressure measurements is systolic blood pressure (SBP) >180 mmHg or diastolic blood pressure (DBP) >100 mmHg
* heart failure NYHA class III or IV
* AST or ALT greater than 3 times the upper limit of normal
* systemic corticosteroids have been used for 10 consecutive days within 90 days (topical, eye drop, topical or inhalation agents)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Glycemic control

SECONDARY OUTCOMES:
Fasting plasma glucose | 6 months
  Glucose metabolism
Postprandial glucose | 6 months
  Glucose metabolism
Whole body muscle | 6 months
  Body composition
Whole body fat | 6 months
  Body composition
Abdominal subcutaneous fat | 6 months
  Body composition
Abdominal visceral fat | 6 months
  Body composition
NTproBNP | 6 months
  Cardiac marker
Troponin T | 6 months
  Cardiac marker
Lipids | 6 months
  Lipid profiles (TG, HDL, and LDL)
Lipoprotein (a) | 6 months
  Lipid metabolism
Urinary microalbumin-Creatinine ratio | 6 months
  Lipid metabolism
Fib-4 | 6 months
  Hepatic fibrosis marker

OTHER OUTCOMES:
Adverse events | 6 months
  Side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided